CLINICAL TRIAL: NCT05203913
Title: Efficacy and Safety of the Combination of Cisplatin Plus Nab-paclitaxel and Nivolumab With Radiotherapy After Maximal Tumor Resection in Non-metastatic Muscle Invasive Bladder Cancer.
Brief Title: Cisplatin, Nab-paclitaxel, Nivolumab With Radiotherapy After Resection of Non-Metastatic Muscle Invasive Bladder Cancer
Acronym: CNN-BC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4353
Record Dates: First submitted 2021-11-29; First posted 2022-01-24 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-09

CONDITIONS: Muscle-Invasive Bladder Carcinoma
Keywords: nivolumab; nab-paclitaxel; cisplatin; trimodal therapy; radiotherapy
MeSH Terms: interventions — Nivolumab; Taxes; Albumin-Bound Paclitaxel; Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental arm (Experimental): This arm consists in treatment with cisplatin + nab-paclitaxel + nivolumab during radiotherapy on bladder followed by nivolumab alone after the end of radiotherapy
  Interventions: Drug: Nivolumab; Drug: Nab paclitaxel; Drug: Cisplatin; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Nivolumab — The recommended dose for nivolumab is 480 mg administered as 30 minutes IV infusions every 28 days for 13 infusions.
  Other Names: Opdivo
Drug: Nab paclitaxel — The recommended dose for nab-paclitaxel is 60 mg per square meter administered as 30 minutes IV infusions every 7 days (weekly), during the radiotherapy period.
  Other Names: Abraxane
Drug: Cisplatin — The recommended dose for cisplatin is 20 mg per square meter administered as 60 minutes IV infusions every 7 days (weekly), during the radiotherapy period.
  Other Names: CDDP
Radiation: Radiotherapy — Radiotherapy will be delivered over approximately 5 weeks.The total radiotherapy dose will be: 60 Gray in 25 fractions over 5 weeks on original bladder tumour, 50 Gray in 25 fractions over 5 weeks on whole bladder and pelvic nodes if included, administered as concomitant boost. Radiation therapy will be delivered once daily (Monday-Friday) continuously without a planned break for tumour response assessment during treatment.
  Other Names: RT

SUMMARY:
In this phase II study, eligible patients will be treated with maximal tumor resection and then started treatment within 8 weeks. Chemotherapy, Nivolumab and radiotherapy (RT) will be started on day one. Chemotherapy will be administered weekly during radiotherapy. Radiotherapy will be performed from Monday to Friday for five weeks. Nivolumab will be administered for one year (13 infusions).

Patients will have the complete tumour assessment by computed tomography scan (CT-scan) and cystoscopy up to 5 years after radiotherapy.

DETAILED DESCRIPTION:
The screening phase is up to six weeks before the beginning of treatment. The treatment phase is from the day one of therapy until 30 days after the last patient last cycle. During the treatment phase each patient will be treated with concomitant chemo-radiotherapy for up to five weeks. The first day of radiotherapy is considered the first day of treatment in the study and cisplatin, nab-paclitaxel and nivolumab will be administered. Cisplatin and nab paclitaxel will be administered weekly during radiotherapy for a maximum of five infusions. Nivolumab will be administered at a flat dose of 480 mg every four weeks for 13 cycles. After the end of radio-chemotherapy patients will be followed every four weeks until the end of nivolumab treatment of up to 13 cycles.

Radiological assessment with whole body (abdominal/pelvic/chest) CT-scan or CT-scan of the thorax and abdominal magnetic resonance imaging (MRI). This will be performed every 16 weeks (±2 weeks) after the post radio/chemotherapy evaluation for the first two years and every six months (±2 weeks) up to 5 years. After five years patients will be followed as per local clinical practice.

At the time of radiographic disease progression, patients exit from the study and will be managed as per local guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old or older
2. Histologic diagnosis of predominantly urothelial carcinoma of the bladder. Focal differentiation allowed other than small cell histology.
3. Stage T2-T3 N0M0 (AJCC-TNM version 6) based on trans-urethral resection of bladder tumor (TURBT), CT or MRI imaging, +/- bimanual examination under anaesthesia.
4. FDG-PET within 6 weeks from the start of treatments, showing no evidence of lymph nodes or metastatic disease.
5. Attempt of complete trans urethral resection of bladder tumour (TURBT) within 56 days (8 weeks) prior to the start of chemoradiotherapy. If TURBT was performed > 8 weeks prior but a recent cystoscopy shows no residual disease, then a repeat TURBT is not necessary.
6. Life expectancy greater than 6 months
7. Eastern Cooperative Oncology Group (ECOG) performance status of 1 or better
8. Another primary cancer is allowed only if treated with curative intent at least 3 years prior to enrolment without evidence of recurrence or if the untreated cancer is clinically indolent (e.g., lower risk prostate cancer).
9. Patients must be considered able to tolerate systemic chemotherapy combined with pelvic intensity-modulated radiation therapy (IMRT) by the joint agreement of the participating radiation oncologist and medical oncologist.
10. Able and willing to give written informed consent.
11. For women of childbearing potential (WOCBP), study participants must use a contraceptive method that is highly effective (with a failure rate of < 1% per year) for at least 5 months after the last dose of study intervention. Men receiving any study drug and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 6 months after the last dose of chemotherapy with cisplatin or nab-paclitaxel.

    The investigator or a designated associate is requested to advise the subject how to achieve an adequate birth control. Adequate contraception is defined in the study as any medically recommend method (or combination of methods) as per standard of care. Acceptable methods are oral contraceptives, hormonal implants, hormonal patches, IDU, Diaphragm with spermicides, cervical cape with spermicide, and condom with spermicide.
12. Adequate bone-marrow, liver, and renal function as assessed by the following laboratory requirements conducted within 7 days of starting the study treatment:
13. Total bilirubin ≤1∙5 × the upper limit of normal (ULN).
14. Alanine aminotransferase and aspartate aminotransferase ≤2 × ULN (≤5 × ULN for patients with liver involvement of their cancer).
15. International normalized ratio (INR) and partial thromboplastin time (PTT) ≤1∙5 × ULN. Subjects who are therapeutically treated with an agent such as warfarin or heparin will be allowed to participate if no prior evidence of an underlying abnormality in coagulation parameters exists. Close monitoring with at least weekly evaluations will be performed until INR and PTT are stable based on a pre-dose measurement as defined by the local standard of care.
16. Platelet count ≥100 000/mm3, haemoglobin >9 g/dl, absolute neutrophil count >1,500/mm3.
17. Alkaline phosphatase limit ≤2∙5 × ULN (≤5 × ULN for patients with liver involvement of their cancer).
18. Creatinine clearance greater than 40 ml/min as evaluated by Cockcroft-Gault formula.

Exclusion Criteria:

1. Prior systemic therapy for other urothelial tumours.
2. Prior RT to the pelvis
3. Treatment with any other investigational agent or participation in another clinical trial with therapeutic intent within 28 days or five half-lives of the drug, whichever is longer, prior to enrolment.
4. Malignancies other than urothelial cancer within 3 years prior to Cycle 1, Day 1:

   1. Patients with localized lower risk prostate cancer (defined as Stage ≤T2b, Gleason score ≤ 7, and PSA at prostate cancer diagnosis ≤ 20 ng/mL [if measured]) treated with radical prostatectomy and without prostate-specific antigen (PSA) recurrence are eligible.
   2. Patients with lower risk prostate cancer (defined as Stage T1/T2a, Gleason score ≤ 7 and PSA ≤ 10 ng/mL) who are treatment-naive and undergoing active surveillance are eligible.
   3. Patients with malignancies of a negligible risk of metastasis or death (e.g., risk of metastasis or death <5% at 5 years) are eligible provided they meet all the following criteria:
   4. Malignancy treated with expected curative intent (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, or ductal carcinoma in situ of the breast treated surgically with curative intent) No evidence of recurrence or metastasis by follow-up imaging and any disease-specific tumor markers.
5. Pre-existing medical conditions precluding treatment (e.g., previous history of immune-related adverse reactions, pneumonitis, colitis, etc.)
6. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
7. History of autoimmune disease, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjogren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis. Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone may be eligible for this study. Patients with controlled Type I diabetes mellitus on a stable dose of insulin regimen may be eligible for this study.
8. Active tuberculosis
9. For women of childbearing potential (WOCBP), study participants must use a contraceptive method that is highly effective (with a failure rate of < 1% per year) for at least 5 months after the last dose of study intervention. Men receiving any study drug and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 6 months after the last dose of chemotherapy with cisplatin or nab-paclitaxel.

   Acceptable methods are oral contraceptives, hormonal implants, hormonal patches, IDU, Diaphragm with spermicides, cervical cape with spermicide, and condom with spermicide.
10. Received prior therapy with an anti-programmed cell death protein 1 (anti-PD-1), anti-PD-L1, anti-programmed cell death-ligand 2 (anti-PD-L2), anti-CD137 (4-1BB ligand, a member of the Tumor Necrosis Factor Receptor [TNFR] family), or anti-Cytotoxic T-lymphocyte-associated antigen-4 (anti-CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
11. Treatment with systemic corticosteroids or other systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks prior to Cycle 1, Day 1, or anticipated requirement for systemic immunosuppressive medications during the trial.
12. Active autoimmune disease that has required systemic treatment in past 2 years.
13. Received or will receive a live vaccine within 4 weeks prior to first dose of study drug except for vaccine against SARS-CoViD2. Influenza vaccination should be given during influenza season only (approximately October through May in the Northern Hemisphere and approximately April through September in the Southern Hemisphere). Patients must agree not to receive live, attenuated influenza vaccine (e.g., FluMist®) within 28 days prior to randomization, during treatment or within 5 months following the last dose of nivolumab.
14. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
15. Active infection requiring IV systemic therapy.
16. Receipt of therapeutic oral or IV antibiotics within 2 weeks prior to Cycle 1, Day 1. Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or to prevent chronic obstructive pulmonary disease exacerbation) are eligible.
17. Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction within the previous 3 months, unstable arrhythmias, or unstable angina. Patients with known coronary artery disease, congestive heart failure not meeting the above criteria, or left ventricular ejection fraction < 50% must be on a stable medical regimen that is optimized in the opinion of the treating physician, in consultation with a cardiologist if appropriate.
18. Major surgical procedure other than for diagnosis within 28 days prior to Cycle 1, Day 1, or anticipation of need for a major surgical procedure during the course of the study
19. Prior allogeneic stem cell or solid organ transplant
20. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications.
21. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies)
22. Patients with active Hepatitis B virus (HBV) or Hepatitis C virus (HCV)
23. Not willing or unable to sign a consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | From the start of therapy up to 5 years.
  Disease-free survival is defined as the rate of survival free of recurrence in pelvic nodes or bladder, or appearance of distant metastasis with data censored at the first sign of disease or second primary tumor, or death.

SECONDARY OUTCOMES:
Rate of patients who require salvage cystectomy. | From the start of therapy up to 5 years.
  This is the number of patients over the total who had cystectomy after the end of study treatment.
Rate of locoregional Disease Free Survival. | From the start of therapy up to 5 years.
  This is the number of patients over the total who had no bladder or pelvic progression of disease.
Median Disease Free Survival. | From the start of therapy up to 5 years.
  This is defined as the time interval from the start of study treatment to the date of radiological or clinical progression or death due to any cause.
Overall survival | From the start of therapy up to 5 years.
  This is defined as the time interval from the start of study treatment to the date of death due to any cause.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 during treatment with nivolumab plus cisplatin and nab-paclitaxel with concomitant RT. | From the start of therapy up to 30 days after the end of radiotherapy.
  This outcome of safety will include adverse events occurred during the treatment with nivolumab plus cisplatin, nab-paclitaxel and radiotherapy. Adverse events will be classified according to CTCAE criteria version 5.0.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 during treatment with nivolumab alone. | From 30 days after the last dose of radiotherapy up to 100 calendar days from the last dose of nivolumab.
  This outcome of safety will include adverse events occurred during the treatment with nivolumab alone after the end of radiotherapy. Adverse events will be classified according to CTCAE criteria version 5.0.
Quality of life assessed by EQ-5D-5L test. | From the start of therapy up to 30 days after the last dose of treatment.
  Quality of life evaluated by this test comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
Quality of life assessed by NFBlSI-18 test. | From the start of therapy up to 30 days after the last dose of treatment.
  This test evaluate the bladder symptoms and quality of life related to these.

OTHER OUTCOMES:
Median Disease Free Survival by PD-L1 expression. | From the start of therapy up to 5 years.
  Patients with or without PD-L1 expression evaluated by Combined Positive Score (CPS) will be compared in terms of median disease free survival. Patients with CPS ≥ 10 will considered positive, the others negative.
Median Disease Free Survival by PI3KCA mutations | From the start of therapy up to 5 years.
  Patients with or without PI3KCA mutation will be compared in terms of median disease free survival.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Iacovelli, MD, PhD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli IRCCS. Largo A. Gemelli 8, 00168 Rome, Italy.
Locations (1):
- Roberto iacovelli, Roma, Italy

IPD SHARING:
Plan to Share IPD: No